CLINICAL TRIAL: NCT02385279
Title: Multicenter Randomized Study of the MiStent Sirolimus Eluting Absorbable Polymer Stent System (MiStent SES) for Revascularization of Coronary Arteries
Brief Title: Study Comparing the MiStent SES Versus the XIENCE EES Stent
Acronym: DESSOLVE III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ECRI bv (Industry)
Collaborators: Micell Technologies (Industry); Stentys (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECRI-005
Record Dates: First submitted 2015-02-17; First posted 2015-03-11 (Estimated); Results first posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2022-07

CONDITIONS: Coronary Stenosis
Keywords: CAD; ACS; All comers; PCI
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MiStent® (Experimental): Percutaneous Coronary Intervention with the MiStent Sirolimus Eluting Absorbable Polymer Coronary Stent. It is a balloon expandable sirolimus eluting stent with an absorbable polymer coating.
  Interventions: Device: MiStent
- XIENCE EES (Active Comparator): Percutaneous Coronary Intervention with the XIENCE EES (Everolimus Eluting) Coronary Stent System. The stents are balloon expandable drug eluting stents using everolimus with a non-erodible or durable polymer coating.
  Interventions: Device: XIENCE EES

INTERVENTIONS:
Device: MiStent — Percutaneous Coronary Intervention
  Arms: MiStent®
Device: XIENCE EES — Percutaneous Coronary Intervention
  Arms: XIENCE EES

SUMMARY:
The primary objective of this study is to compare the performance of MISTENT to that of XIENCE in an all-comers patient population with symptomatic ischemic heart disease. The patients will be followed through 3 years for major clinical events.

ELIGIBILITY:
Inclusion Criteria:

All comers" patients:

* Male or female patients 18 years or older;
* Presence of one or more coronary artery stenoses of 50% or more in a native coronary artery or in a saphenous venous or arterial bypass conduit suitable for coronary stent implantation.
* The vessel should have a reference vessel diameter ranging from 2.5 mm to 3.75 mm (no limitation on the number of treated lesions, vessels, or lesion length); All lesions of the patient must comply with the angiographic inclusion criteria.
* The patient is judged to be capable of providing voluntary informed consent and has been fully informed of the nature of the study, is willing to comply with all study requirements and will provide written informed consent as approved by the Ethics Committee of the respective clinical site.

Exclusion Criteria:

* Known pregnancy or breastfeeding at time of randomization;
* Known contraindication or hypersensitivity to sirolimus, everolimus, cobalt-chromium, or to medications such as aspirin, heparin, bivalirudin, and all of the following four medications: clopidogrel bisulfate, ticlopidine, prasugrel, ticagrelor;
* Concurrent medical condition with a life expectancy of less than 12 months.
* The patient is unwilling/ not able to return for outpatient clinic at 1 month and 12 months follow-up.
* Currently participating in another trial and not yet at its primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1398 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Spitzer, MD, Study Director — European Cardiovascular Research Institute
Locations (20):
- France (3):
  - Research Center Corbeil, Corbeil
  - Research Center Nimes, Nîmes
  - Research Center Poitiers, Poitiers
- Germany (5):
  - Research Center Jena, Jena
  - Research Center Leipzig, Leipzig
  - Research Center Munster, Münster
  - Research Center Ulm, Ulm
  - Research Center Wiesbaden, Wiesbaden
- Netherlands (7):
  - Research Center Amersfoort, Amersfoort
  - Research Center Amsterdam, Amsterdam
  - Tergooi, Blaricum
  - Research Center Emmen, Emmen
  - Research Center Leeuwarden, Leeuwarden
  - Research Center Nijmegen, Nijmegen
  - Research Center Venlo, Venlo
- Poland (5):
  - Research Center Belchatow, Bełchatów
  - Research Center Bielsko-Biala, Bielsko-Biala
  - Research center Chrzanow, Chrzanów
  - Research Center Tychy, Tychy
  - Research Center Zgierz, Zgierz

REFERENCES:
- [Background] de Winter RJ, Katagiri Y, Asano T, Milewski KP, Lurz P, Buszman P, Jessurun GAJ, Koch KT, Troquay RPT, Hamer BJB, Ophuis TO, Wohrle J, Wyderka R, Cayla G, Hofma SH, Levesque S, Zurakowski A, Fischer D, Kosmider M, Goube P, Arkenbout EK, Noutsias M, Ferrari MW, Onuma Y, Wijns W, Serruys PW. A sirolimus-eluting bioabsorbable polymer-coated stent (MiStent) versus an everolimus-eluting durable polymer stent (Xience) after percutaneous coronary intervention (DESSOLVE III): a randomised, single-blind, multicentre, non-inferiority, phase 3 trial. Lancet. 2018 Feb 3;391(10119):431-440. doi: 10.1016/S0140-6736(17)33103-3. Epub 2017 Dec 5. PMID 29203070
- [Derived] Wang R, Kawashima H, Hara H, Gao C, Ono M, Takahashi K, Tu S, Soliman O, Garg S, van Geuns RJ, Tao L, Wijns W, Onuma Y, Serruys PW. Comparison of Clinically Adjudicated Versus Flow-Based Adjudication of Revascularization Events in Randomized Controlled Trials. Circ Cardiovasc Qual Outcomes. 2021 Nov;14(11):e008055. doi: 10.1161/CIRCOUTCOMES.121.008055. Epub 2021 Oct 20. PMID 34666500
- [Derived] Katagiri Y, Andreini D, Miyazaki Y, Takahashi K, Komiyama H, Mushtaq S, Sonck J, Schoors D, Maisano F, Kaufman PA, Leal I, Lindeboom W, Piek JJ, Wykrzykowska JJ, Morel MA, Bartorelli AL, Onuma Y, Serruys PW; SYNTAX III REVOLUTION Investigators. Site vs. core laboratory variability in computed tomographic angiography-derived SYNTAX scores in the SYNTAX III trial. Eur Heart J Cardiovasc Imaging. 2021 Aug 14;22(9):1063-1071. doi: 10.1093/ehjci/jeaa172. PMID 32888011
- [Derived] Takahashi K, Serruys PW, Kogame N, Buszman P, Lurz P, Jessurun GAJ, Koch KT, Troquay RPT, Hamer BJB, Oude Ophuis T, Milewski KP, Hofma SH, Wykrzykowska JJ, Onuma Y, de Winter RJ, Wijns W. Final 3-Year Outcomes of MiStent Biodegradable Polymer Crystalline Sirolimus-Eluting Stent Versus Xience Permanent Polymer Everolimus-Eluting Stent: Insights From the DESSOLVE III All-Comers Randomized Trial. Circ Cardiovasc Interv. 2020 Jun;13(6):e008737. doi: 10.1161/CIRCINTERVENTIONS.119.008737. Epub 2020 May 29. PMID 32466676

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MiStent® | XIENCE EES
Started | 703 | 695
Completed | 676 | 677
Not Completed | 27 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MiStent® | XIENCE EES | Total
Number analyzed (Participants) | 703 | 695 | 1398
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 257 | 271 | 528
  >=65 years | 446 | 424 | 870
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (10.7) | 66.3 (10.7) | 66.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209 | 182 | 391
  Male | 494 | 513 | 1007
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 297 | 296 | 593
  Poland | 187 | 184 | 371
  France | 56 | 56 | 112
  Germany | 163 | 159 | 322

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Occurrence of a Device Oriented Composite Endpoint (DOCE)
Description: DOCE is a composite of clinical endpoint of cardiac death, myocardial infarction not clearly attributable to a non-target vessel and clinically-indicated target lesion revascularization.
Time Frame: 12 months postprocedure
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | MiStent® | XIENCE EES
Number analyzed (Participants) | 703 | 695
Participants | 40 | 45

2. Secondary Outcome: POCE
Description: POCE defined as all-cause death, any Myocardial Infarction (MI), or any revascularization
Time Frame: At 12 months
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | MiStent® | XIENCE EES
Number analyzed (Participants) | 703 | 695
Participants | 93 | 101

3. Secondary Outcome: MACE
Description: MACE defined as all-cause death, any MI, or any Target Vessel Revascularization (TVR)
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MiStent® | XIENCE EES
Number analyzed (Participants) | 703 | 695
Participants | 65 | 65

4. Secondary Outcome: Target Vessel Failure (TVF)
Description: Target Vessel Failure (TVF) defined as cardiac death, TV MI, or clinically indicated TVR
Time Frame: At 12 months
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | MiStent® | XIENCE EES
Number analyzed (Participants) | 703 | 695
Participants | 45 | 53

5. Secondary Outcome: All-cause Death
Description: All-cause death
Time Frame: At 12 months
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | MiStent® | XIENCE EES
Number analyzed (Participants) | 703 | 695
Participants | 25 | 18

6. Secondary Outcome: Myocardial Infarction
Description: Any Myocardial infarction
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MiStent® | XIENCE EES
Number analyzed (Participants) | 703 | 695
Participants | 17 | 15

7. Secondary Outcome: Any Revascularization
Description: Any revascularization
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MiStent® | XIENCE EES
Number analyzed (Participants) | 703 | 695
Participants | 61 | 78

8. Secondary Outcome: Stent Thrombosis
Description: Definite or probably stent thrombosis according to ARC
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MiStent® | XIENCE EES
Number analyzed (Participants) | 703 | 695
Participants | 5 | 6

ADVERSE EVENTS:
Time Frame: 12 months (primary reporting), and yearly up to 5 years.
Description: Adverse event reporting in the context of a post-marketing trial.
Arm/Group | MiStent® | XIENCE EES
All-Cause Mortality (participants affected / at risk) | 85/703 | 78/695
Serious Adverse Events (participants affected / at risk) | 434/703 | 426/695
Other Adverse Events (participants affected / at risk) | 76/703 | 71/695
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MiStent® (N=703) | XIENCE EES (N=695)
Myocardial infarction (Cardiac disorders) | 17 | 15
Definite stent thrombosis (Cardiac disorders) | 3 | 5
Other (General disorders) | 414 | 406
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MiStent® (N=703) | XIENCE EES (N=695)
Non Serious AE (General disorders) | 76 | 71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/79/NCT02385279/Prot_SAP_000.pdf